CLINICAL TRIAL: NCT01959490
Title: Next Generation Sequencing to Evaluate Breast Cancer Subtypes and Genomic Predictors of Response to Therapy in the Preoperative Setting for Stage II-III Breast Cancer
Brief Title: Trastuzumab and Pertuzumab or Bevacizumab With Combination Chemotherapy in Treating Patients With Stage II-III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CASE14112; NCI-2013-01422 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 14112 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2013-08-16; First posted 2013-10-10 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; pertuzumab; Docetaxel; Carboplatin; Doxorubicin; Cyclophosphamide; Paclitaxel; Taxes; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1P (HER2 positive) (Experimental): Patients receive a run-in Pertuzumab treatment of 840 mg IV over 60 minutes on day -14 followed by Trastuzumab IV over 30-60 minutes and Pertuzumab IV over 30-60 minutes, docetaxel IV, and carboplatin IV on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Biological: Pertuzumab; Drug: docetaxel; Drug: carboplatin
- Cohort 1T (HER2 positive) (Experimental): Patients receive a run-in Trastuzumab treatment of 8 mg/kg IV over 90 minutes on day -14 followed by Trastuzumab IV over 30-60 minutes and Pertuzumab IV over 30-60 minutes, Docetaxel IV, and Carboplatin IV on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Biological: Pertuzumab; Drug: docetaxel; Drug: carboplatin
- Cohort II (HER2 negative) (Experimental): Patients receive Bevacizumab IV over 30-60 minutes on day 1 of weeks 1, 3, 5, 7, 9, and 11; Doxorubicin IV and Cyclophosphamide IV over 30-60 minutes on day 1 of weeks 1, 3, 5, and 7; and Paclitaxel IV over 3 hours on day 1 of weeks 9, 11, 13, and 15.
  Interventions: Drug: doxorubicin; Drug: cyclophosphamide; Drug: paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
  Arms: Cohort 1P (HER2 positive); Cohort 1T (HER2 positive)
Biological: Pertuzumab — Given IV
  Other Names: 2C4; Perjeta
  Arms: Cohort 1P (HER2 positive); Cohort 1T (HER2 positive)
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
  Arms: Cohort 1P (HER2 positive); Cohort 1T (HER2 positive)
Drug: carboplatin — Given IV
  Other Names: Carboplat; CBDCA; JM-8; Paraplat; Paraplatin
  Arms: Cohort 1P (HER2 positive); Cohort 1T (HER2 positive)
Drug: doxorubicin — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF; doxorubicin hydrochloride
  Arms: Cohort II (HER2 negative)
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
  Arms: Cohort II (HER2 negative)
Drug: paclitaxel — Given IV
  Other Names: Anzatax; Asotax; TAX; Taxol
  Arms: Cohort II (HER2 negative)
Drug: Bevacizumab
  Other Names: Avastin
  Arms: Cohort II (HER2 negative)

SUMMARY:
This phase II trial studies how well trastuzumab and pertuzumab or bevacizumab with combination chemotherapy works in treating patients with stage II-III breast cancer. Monoclonal antibodies, such as trastuzumab, pertuzumab, and bevacizumab, can block tumor growth in different ways. Some block the ability of tumors to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as docetaxel, carboplatin, doxorubicin hydrochloride, cyclophosphamide, and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving trastuzumab and pertuzumab or a commercially marketed formulation of bevacizumab without modification with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if genomically derived 'molecular subtypes' predict pathological complete response to combination chemotherapy and targeted therapy for HER2 early stage breast cancer.

SECONDARY OBJECTIVES:

I. To explore the ability of trastuzumab or pertuzumab response signatures to predict pCR in HER2 positive tumors treated with brief exposure to trastuzumab or pertuzumab followed by combination chemotherapy.

II. To explore the value of immune signatures as well as AKT and IGF signatures to predict pCR in HER2 tumors treated with brief exposure to trastuzumab and pertuzumab.

III. To explore if comprehensive annotation of genomic alterations (mutations, copy number alternations, gene fusions, non-coding RNA and splice variants) can further sub-stratify subtype-based classifiers for prediction of response to targeted therapy in early stage breast cancer IV. To explore if circulating RNA expression levels are associated with treatment response V. To explore changes in cardiac function and identify early cardiac injury using strain echocardiograms and cardiac biomarkers during treatment VI. To explore immunohistochemistry-based markers of response to treatment

Objectives for Imaging Sub-Study: Secondary Objectives I. Evaluate the visualization of primary breast tumors using analog and digital positron emission tomography (PET) with FDG and FLT. II. Evaluate the quantification of FDG-uptake in primary breast tumors using analog and digital PET with FDG and FLT. III. Compare the levels and changes in metabolic tumor activity from analog and digital FDG-PET/CT or FLT-PET/CT with clinical follow up and other procures include into CASE 14112 (such as DCE-MRI, genetic testing, etc.)

OUTLINE: Patients are assigned to 1 of 2 treatment cohorts based on HER2 status.

COHORT I (HER2 positive): Patients receive trastuzumab intravenously (IV) over 30-60 minutes, and pertuzumab IV over 30-60 minutes, docetaxel IV, and carboplatin IV on day 1. Treatment repeats every 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity. As part of standard of care, each patient will receive three MRIs pre-treatment, before biopsy is taken, and before surgery. Ten additional patients will be added to cohort 1 to take part in the imaging sub-study. These ten patients will follow the same procedure as the other participants in cohort I but will have a PET/CT in place of the DCE-MRI

COHORT II (HER2 negative): Patients receive bevacizumab IV over 30-60 minutes on day 1 of weeks 1, 3, 5, 7, 9, and 11; doxorubicin IV and cyclophosphamide IV over 30-60 minutes on day 1 of weeks 1, 3, 5, and 7; and paclitaxel IV over 3 hours on day 1 of weeks 9, 11, 13, and 15. Prior to receiving paclitaxel patients will receive the anti-nausea medication

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the breast, with sufficient tissue available for estrogen receptor (ER), progesterone receptor (PR), and HER 2 testing

  * HER2 must be positive by IHC or ISH testing by laboratory standard.
* Needle biopsy or incisional biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Resectable disease-clinical stage I (T/0/N0miT1N0-N0mi), IIA-IIIA (T2 N0/T3N0 or T1-3 N1-N2a) or unresectable disease - clinical stage IIIB/IIIC (T4 or T1-3 N2b-3); no evidence of metastatic disease
* No prior chemotherapy, hormonal therapy, or radiation therapy for this cancer
* Absolute neutrophil count (ANC) ≥1000/ul
* Platelet count ≥ 100,000/ul
* Hemoglobin ≥ 9 g/dl
* Serum creatinine ≤ 1.5 mg/dl or measured creatinine clearance of > 30 ml/min
* Total bilirubin ≤ upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 x ULN
* Patients with multiple foci of invasive cancer in the same breast are eligible if any single lesion meets the above size criteria and all sampled lesions are histologically similar (whether radiographically detected lesions separate from the target lesion are sampled for histologic evaluation is left to the discretion of the treating physicians); the presence of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS) in either breast will not render a patient ineligible; patients with a small focus of invasive cancer detected the contralateral breast (clinical T1N0) are eligible, however only the histologic response in the breast containing the target lesions will be considered in determining the patient's pathologic response
* Measurable disease in the breast or axilla that measures at least 1 cm by either clinical or radiographic measurement

Exclusion Criteria:

* Excisional biopsy
* Pregnant and lactating women are not eligible; all participants of reproductive age must have a negative serum pregnancy test at baseline and agree to use an effective barrier method of contraception during the entire period of treatment on the study
* Patients with New York Heart Association (NYHA) grade 2 or higher congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, or arterial thrombotic event with the past 12 months, uncontrolled hypertension (systolic blood pressure > 150 and/or diastolic blood pressure > 100 on antihypertensive medications; patients not on medication for high blood pressure who are found to have systolic blood pressure [SBP] > 150 and/or diastolic blood pressure [DBP] > 100 should have 3 documented episodes of elevated blood pressure before being considered 'uncontrolled', if they have 3 documented episodes of elevated blood pressure, then can be started on antihypertensive medications; patients currently on antihypertensive medications with elevated blood pressures as defined above may have their medications adjusted; if patients have persistent [3 episodes] of high blood pressure despite medication adjustment they will be considered ineligible for study participation; each measured episode should be 24 hours apart), prior history of hypertensive crisis or hypertensive encephalopathy, uncontrolled or clinically significant arrhythmia, grade II or greater peripheral vascular disease or prior history of stroke or transient ischemic attack (TIA); patient must have a pretreatment multi gated acquisition scan (MUGA) scan or echocardiogram with left ventricular ejection fraction (LVEF) above lower limit of normal
* No non-breast malignancy within the past 5 years other than treated squamous or basal cell carcinoma of the skin or CIS of the cervix
* Patients known to be human immunodeficiency virus (HIV) positive are not eligible for the study given their potentially compromised immune systems and increased risk of treatment-related toxicity
* Advanced (T1N1-4/T2-3 N any) invasive cancer in the contralateral breast
* Any known history of cerebrovascular disease including TIA, stroke or subarachnoid hemorrhage
* Patients must not have a non-healing wound or fracture
* Patients with an abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months
* Patients must not have a bleeding diathesis, hereditary of acquired bleeding disorder or coagulopathy
* Patients on therapeutic doses of Coumadin or Lovenox are ineligible to participate in study
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study; core biopsy or other minor surgical procedure, for example placement of a vascular access device, are excluded from this requirement
* No known hypersensitivity to any component of bevacizumab

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-09-24 (Actual); Primary Completion 2016-11-11 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Silverman, MD, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1P (HER2 Positive): Patients receive a run-in Pertuzumab treatment of 840 mg IV over 60 minutes on day -14 followed by Trastuzumab IV over 30-60 minutes and Pertuzumab IV over 30-60 minutes, docetaxel IV, and carboplatin IV on day 1. Treatment repeats very 3 weeks for 6 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Started | 5 | 6 | 5
Completed | 5 | 6 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants enrolled in study
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative) | Total
Number analyzed (Participants) | 5 | 6 | 5 | 16
Age, Customized [Count of Participants; unit: Participants]
  30-39 years | 0 | 1 | 0 | 1
  40-49 years | 1 | 2 | 1 | 4
  50-59 years | 3 | 1 | 0 | 4
  60-69 years | 0 | 1 | 4 | 5
  70-79 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 5 | 16
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 5 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 0 | 3
  White | 4 | 4 | 5 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Pathological Complete Response (pCR) Who Received Targeted Therapy With Trastuzumab and Pertuzumab or Bevacizumab Predicted by Genomically-derived Molecular Subtypes.
Description: Number of patients with a pathological complete response (pCR) who received targeted therapy with trastuzumab and pertuzumab or bevacizumab predicted by genomically-derived molecular subtypes (HER2 positive or HER2 negative. pCR is defined as absence of invasive cancer in breast or lymph nodes after neoadjuvant chemotherapy.
Time Frame: Up to 30 days after last cycle of treatment
Population: All participants enrolled in study and who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Number analyzed (Participants) | 5 | 6 | 5
Participants | 4 | 6 | 3

2. Secondary Outcome: The Number of HER2 Positive Patients With a Pathological Complete Response (pCR) Predicted by a Trastuzumab and Pertuzumab Response Signature
Time Frame: Up to 30 days after last cycle of treatment
Population: Data not collected
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: The Number of HER2 Negative Patients With a pCR Predicted by the TGF-B Response Signature
Time Frame: Up to 30 days after last cycle of treatment
Population: Data not collected
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: The Number of HER2 Positive Patients With a pCR Predicted by the AKT Signature and IGF Signature.
Time Frame: Up to 30 days after last cycle of treatment
Population: Data not collected
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: The Number of Patients With a pCR Predicated by Copy Number Alterations.
Time Frame: Up to 30 days after last cycle of treatment
Population: Data not collected
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: The Number of Patients With a pCR Predicted by Changes in Texture on Breast DCE-MRI After a Two-week "run-in" Treatment With Trastuzumab, Pertuzumab, or Bevacizumab
Description: Determine if changes in regularity and entropy range predict pCR and in an exploratory fashion determine if specific texture features exist in each molecular subtype that predict pCR.
Time Frame: At 2 weeks after start of run-in period
Population: Data not collected
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Number analyzed (Participants) | 0 | 0 | 0

7. Other Pre Specified Outcome: Descriptive Statistics of PET/CT Scan
Description: Qualitative and quantitative image analysis will be performed and descriptively summarized. For the 10 patients in the PET/CT sub-study of cohort 1.
Time Frame: Up to 30 days after last cycle of treatment
Population: Outcome not determined because low accrual prevented appropriate analysis and calculation of the prediction measure.
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last cycle of treatment
Arm/Group | Cohort 1P (HER2 Positive) | Cohort 1T (HER2 Positive) | Cohort II (HER2 Negative)
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/6 | 1/5
Other Adverse Events (participants affected / at risk) | 5/5 | 3/6 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1P (HER2 Positive) (N=5) | Cohort 1T (HER2 Positive) (N=6) | Cohort II (HER2 Negative) (N=5)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1P (HER2 Positive) (N=5) | Cohort 1T (HER2 Positive) (N=6) | Cohort II (HER2 Negative) (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (8) | 3 (6) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 2 (2) | 2 (7)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes